CLINICAL TRIAL: NCT03708874
Title: Comparison of Intravenous Paracetamol and Intraperitoneal Bupivacaine for Acute Laparoscopic Cholecystectomy Pain Relief in Patients With Acute Cholecystitis. A Prospective Randomized Clinical Trial
Brief Title: Pain Management of Emergency Laparoscopic Cholecystectomy in Patients With Acute Cholecystitis
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Turgut Donmez, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: BakirköyEAH 2
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Abdominal Pain; Shoulder Pain; Satisfaction; Complication
MeSH Terms: conditions — Abdominal Pain; Shoulder Pain; Personal Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1.Intraoperative bupivacaine: intraperitoneal bupivacaine wash-emergency laparoscopic cholecystectomy
- Group 2.Intravenous paracetamol: intravenous paracetamol-emergency laparoscopic cholecystectomy

SUMMARY:
Patients diagnosed with acute cholecystitis benefit from emergency laparoscopic cholecystectomy (LC). Patients who had emergency LC showed improvement in quality of life in one month compared to those treated. Delayed LC (after the acute cholecystitis has passed) and less time to recover from work. This strategy reduces the risk of repeated referrals with more pain or pancreatitis. There are many studies on the efficacy of intraoperative intraperitoneal bupivacaine(IPBV) with elective LC on pain of IPBV. However, the prospective study of reducing the postoperative pain of emergency LC - IPBV is very few. This study will be conducted to evaluate the efficacy of IPBV in patients with emergency LC.

DETAILED DESCRIPTION:
Patients to be included in the study will be selected from the group between 18 and 70 years of age who apply to general surgery and emergency policlinics, depending on patient approval. All patients will be informed about the operation and the procedures to be performed. Patients who accepted to participate in the study will be included in the study and randomization will be performed by randomly selected patients and two groups. The study will be carried out by 2 surgeons with 5 years of laparoscopic cholecystectomy (LC).Adult patients presenting with acute cholecystitis treated by emergency surgeons by one of two surgeons will be included in the study. These two surgeons will be responsible for the participant records. 1.hepatobiliary ultrasound-confirmed acute cholecystitis diagnosis, 2. Patients undergoing elective laparoscopic cholecystectomy (el-LC) will not be included in the study. Patients converted into an open procedure will be excluded from the study. Patients will be divided into two groups. In Group A, intravenous 1 gr paracetamol via will be applied in 30 minutes after waking up.In Group B, immediately after the introduction of intraoperative laparoscopic trocars, 480 ml of saline + 20 ml of 5% bupivacaine solution will be washed in the subdiaphragmatic area, gallbladder region and the entire abdomen. In both groups, standard laparoscopic cholecystectomy will be performed. In both groups, nasogastric tube will be inserted at the end of the operation after intubation. , CRP(C-reactive protein) levels, ALT(Alanine Aminotransferase) , AST(Aspartate Aminotransferase), GGT(Gamma-Glutamyltransferase), total bilirubin, direct bilirubin values will be recorded. Pulse, heart rate, systolic and diastolic pressures, Oxygen saturation (with pulse) during surgery will be recorded in both groups. Post-operative VAS(Visual analogue score) and VRS(Verbal Rating Scales) pain scores will be performed. VAS 0-10 cm and VRS (no pain in cough (score = 0); pain in cough, not in deep breathing (score = 1); resting (score = 2), pain at rest, mild (score = 3); pain at rest, severe (score = 4)) will be evaluated as.

ELIGIBILITY:
Inclusion Criteria:

* Acute stone cholecystitis
* Acute acrylic cholecystitis

Exclusion Criteria:

* Cholecystitis with chronic stones
* Gallbladder polyps,
* Patients with bleeding diathesis,
* Allergy to local anesthetic agents,
* Patients with paracetamol group allergy,
* Choledocholithiasis associated with acute cholecystitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 18-70 years diagnosed with ASA I, II and III acute cholecystitis
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Post-operative Shoulder Pain | postoperative 1st day
  Group 1 and Group 2 Post-operative shoulder pain. VAS score ;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.

SECONDARY OUTCOMES:
Post-operative Abdominal Pain 2nd Hour | pain at postoperative 2nd hour
  VAS score ;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.
operation time | up to 100 minutes
  duration of operation(minutes), time from anesthesia induction to extubation of the patient
Change in C -reactive protein (CRP) level in all study participants | preoperative and postoperative 1st day
  Compare the postoperative 1st day CRP levels with the baseline CRP in study patients. Comparison will be performed using a paired t-test.
Change in alanine aminotransferase (ALT) level in all study participants | preoperative and postoperative 1st day
  Compare the postoperative 1st day ALT levels with the baseline ALT in study patients. Comparison will be performed using a paired t-test.
Change in Aspartate Aminotransferase (AST) level in all study participants | preoperative and postoperative 1st day
  Compare the postoperative 1st day AST levels with the baseline AST in study patients. Comparison will be performed using a paired t-test.
Post-operative Abdominal Pain 6th Hour | pain at postoperative 6th hour
  VAS score ;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.
Post-operative Abdominal Pain 12th Hour | pain at postoperative 12th hour
  VAS score ;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.
Post-operative Abdominal Pain 24th Hour | pain at postoperative 24th hour
  VAS score ;Explain to the person that each number describe the intensity of his pain. Number 0 describe very happy and no pain and no hurt at all. Number 1 hurts just a little bit. And as te numbers gradually increase pain will increase. Number 10 describes the worst pain in his life. Ask the patient to choose the number that best describes how he is feeling and his pain.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Donmez, surgeon, Principal Investigator — Bakirkoy Training and Research Hospital; Mehmet Emin Gunes, MD, Study Director — Bakirkoy Training and Research Hospital
Locations (1):
- Turgut Donmez, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the patients are included in the study, the patient data will be entered into the system and the results will be evaluated.

REFERENCES:
- [Result] Gurusamy KS, Nagendran M, Toon CD, Guerrini GP, Zinnuroglu M, Davidson BR. Methods of intraperitoneal local anaesthetic instillation for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 25;2014(3):CD009060. doi: 10.1002/14651858.CD009060.pub2. PMID 24668032
- [Result] Kaushal-Deep SM, Anees A, Khan S, Khan MA, Lodhi M. Randomized controlled study of intraincisional infiltration versus intraperitoneal instillation of standardized dose of ropivacaine 0.2% in post-laparoscopic cholecystectomy pain: Do we really need high doses of local anesthetics-time to rethink! Surg Endosc. 2018 Jul;32(7):3321-3341. doi: 10.1007/s00464-018-6053-z. Epub 2018 Jan 16. PMID 29340809
- [Result] Roberts KJ, Gilmour J, Pande R, Hodson J, Lam FT, Khan S. Double-blind randomized sham controlled trial of intraperitoneal bupivacaine during emergency laparoscopic cholecystectomy. Hepatobiliary Pancreat Dis Int. 2013 Jun;12(3):310-6. doi: 10.1016/s1499-3872(13)60049-1. PMID 23742777